CLINICAL TRIAL: NCT03621553
Title: Vitamin D Homeostasis in Sarcoidosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Connie C W Hsia, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU 062010-055
Record Dates: First submitted 2018-07-17; First posted 2018-08-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Sarcoidosis; Vitamin D Insufficiency
MeSH Terms: conditions — Sarcoidosis | interventions — Ergocalciferols; Calcium Citrate

STUDY DESIGN:
Intervention Model Description: Vitamin-D insufficient subjects will receive either vitamin D2 repletion or placebo Vitamin-D sufficient subjects will be observed without treatment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Groups separated by a) use / non-use of oral prednisone, and b) status of serum 25-hydroxy-vitamin-D level (sufficient or insufficient). Those who are vitamin-D insufficient will be randomized to receive either vitamin D2 or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Low vit-D, Ergocalciferol (Experimental): Low serum vitamin D level, split by use or non-use of systemic corticosteroid. Vitamin D2 (Ergocalciferol) 50,000 units will be given by mouth once a week for 12 weeks, then once a month for 12 weeks.
  Daily dietary requirement (calcium citrate with vitamin D2 (200 mg/250 Units tablets, 4 tablets per day) will be given by mouth for 24 weeks).
  Interventions: Drug: Ergocalciferol; Drug: Calcium Citrate with Vitamin D2
- Low vit-D, Placebo (Placebo Comparator): Low serum vitamin D level, split by use or non-use of systemic corticosteroid. Placebo capsules of identical size and appearance will be given by mouth once a week for 12 weeks, then once a month for 12 weeks.
  Daily dietary requirement (calcium citrate with vitamin D2 (200 mg/250 Units tablets, 4 tablets per day) will be given by mouth for 24 weeks).
  Interventions: Drug: Placebo; Drug: Calcium Citrate with Vitamin D2
- Normal vit-D, control (Other): Normal serum vitamin D level, split by use or non-use of systemic corticosteroid.
  Daily dietary requirement (calcium citrate with vitamin D2 (200 mg/250 Units tablets, 4 tablets per day) will be given by mouth for 24 weeks).
  Interventions: Drug: Calcium Citrate with Vitamin D2

INTERVENTIONS:
Drug: Ergocalciferol — Vitamin D2 50,000 units
  Other Names: Vitamin D2
  Arms: Low vit-D, Ergocalciferol
Drug: Placebo — Sugar pill manufactured to mimic ergocalciferol 50,000 units
  Other Names: Placebo oral tablets
  Arms: Low vit-D, Placebo
Drug: Calcium Citrate with Vitamin D2 — To meet the recommended minimum daily dietary requirements
  Other Names: Citracal

SUMMARY:
This study evaluates the relationship between vitamin-D status and severity of sarcoidosis, and the effects of vitamin-D repletion in vitamin-D insufficient patients with sarcoidosis. Half the patients with sarcoidosis who are vitamin-D insufficient will receive standard vitamin-D supplementation via standard regimen while the other half will receive a placebo. Sarcoidosis patients who are vitamin-D sufficient will also act as controls.

DETAILED DESCRIPTION:
Sarcoidosis is a multi-system inflammatory disease characterized by T-helper lymphocyte hyperactivity leading to granulomatous inflammation. The granuloma cells autonomously convert 25-hydroxy-vitamin-D (25OHD) to the active metabolite 1,25-dihydroxy-vitamin-D (1,25OH2D) independent of normal feedback control but dependent on substrate (25OHD) concentration.

Circulating 1,25OH2D exerts both anti-inflammatory and mineral metabolic actions. Deficiency of 25OHD limits substrate-dependent 1,25OH2D synthesis, diminishes anti-antigenic innate immunity and augments pro-inflammatory adaptive immunity. Thus, low vitamin-D stores could aggravate sarcoid inflammation while repletion of vitamin-D stores could mitigate inflammation in sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

* Stable medical condition defined as no hospitalization or emergency room visit in the previous 3 months
* No evidence of active pulmonary or systemic infection
* No other active inflammatory disease,
* No active malignancy.
* Normal serum ionized calcium level

Exclusion Criteria:

* Hospitalization or emergency room visit in the previous 3 months
* Evidence of active pulmonary or systemic infection
* Evidence of active other inflammatory disease
* Evidence of active malignancy
* Elevated serum ionized calcium level

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-07-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in lung function from baseline | Baseline and 24 weeks
  (Measurement at end of study)/(measurement at enrollment)

SECONDARY OUTCOMES:
Change in King's Sarcoidosis Questionnaire Score | Baseline, 12 and 24 weeks
  Standard validated questionnaire for assessing the impact of sarcoidosis on quality of life. Questions address symptoms, activities and psychosocial impacts of disease. It consists of 29 questions on general health, medications, and symptoms in lung, skin, and eyes, summed to derive a total score. Each question is scored on a scale of 1 (worst) to 7 (best). Minimum total score = 5 (poorest health). Maximum total score = 203 (best health).
Change in six minute walk distance | Baseline and 24 weeks
  (Measurement at end of study)/(measurement at enrollment)
Change in blood cell counts from complete blood count (CBC) | Baseline, 12 and 24 weeks
  (Measurement at study point)/(initial measurement at enrollment)
Change in metabolic profile from complete metabolic panel (CMP) | Baseline, 12 and 24 weeks
  (Measurement at study point)/(initial measurement at enrollment)
Change in serum vitamin-D metabolite concentration | Baseline, 12 and 24 weeks
  (Measurement at study point)/(initial measurement at enrollment)
Change in serum angiotensin converting enzyme (ACE) concentration | Baseline, 12 and 24 weeks
  (Measurement at study point)/(initial measurement at enrollment)
Change in serum serum gamma-globulin concentration | Baseline, 12 and 24 weeks
  (Measurement at study point)/(initial measurement at enrollment)
Change in serum C-reactive protein (CRP) concentration | Baseline, 12 and 24 weeks
  (Measurement at study point)/(initial measurement at enrollment)
Change in serum tumor Necrosis factor-alpha (TNF-alpha) concentration | Baseline, 12 and 24 weeks
  (Measurement at study point)/(initial measurement at enrollment)
Change in serum interferon-gamma (IFN-gamma) concentration | Baseline, 12 and 24 weeks
  (Measurement at study point)/(initial measurement at enrollment)
Changes in serum interleukin concentration | Baseline, 12 and 24 weeks
  (Measurement at study point)/(initial measurement at enrollment)
Change in 24 hour urine calcium/creatinine ratio | Baseline, 12 and 24 weeks
  (Measurement at study point)/(initial measurement at enrollment)
Change in 24 hour urine deoxypyridinoline concentration | Baseline, 12 and 24 weeks
  (Measurement at study point)/(initial measurement at enrollment)
Change in fractional lung tissue volume on computed/positron emission tomography (PET/CT) | Baseline and 24 weeks
  (Measurement at end of study)/(measurement at enrollment)
Change in Fluoro-deoxyglucose (FDG) uptake on PET/CT | Baseline and 24 weeks
  (Measurement at end of study)/(measurement at enrollment
Change in bone density z-score | Baseline and 24 weeks
  (Measurement at end of study)/(measurement at enrollment)

CONTACTS AND LOCATIONS:
Overall Officials: Connie Hsia, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, and Parkland Health and Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Result] Capolongo G, Xu LH, Accardo M, Sanduzzi A, Stanziola AA, Colao A, Agostini C, Zacchia M, Capasso G, Adams-Huet B, Moe OW, Maalouf NM, Sakhaee K, Hsia CC. Vitamin-D status and mineral metabolism in two ethnic populations with sarcoidosis. J Investig Med. 2016 Jun;64(5):1025-34. doi: 10.1136/jim-2016-000101. Epub 2016 Apr 6. PMID 27053725
- [Result] Vieth R. Why the optimal requirement for Vitamin D3 is probably much higher than what is officially recommended for adults. J Steroid Biochem Mol Biol. 2004 May;89-90(1-5):575-9. doi: 10.1016/j.jsbmb.2004.03.038. PMID 15225842
- [Result] Bolland MJ, Wilsher ML, Grey A, Horne AM, Fenwick S, Gamble GD, Reid IR. Randomised controlled trial of vitamin D supplementation in sarcoidosis. BMJ Open. 2013 Oct 23;3(10):e003562. doi: 10.1136/bmjopen-2013-003562. PMID 24157819
- [Result] Kamphuis LS, Bonte-Mineur F, van Laar JA, van Hagen PM, van Daele PL. Calcium and vitamin D in sarcoidosis: is supplementation safe? J Bone Miner Res. 2014 Nov;29(11):2498-503. doi: 10.1002/jbmr.2262. PMID 24753153